CLINICAL TRIAL: NCT00689325
Title: A Non-interventional Study Evaluating Well-being/Quality of Life in Schizophrenic Patients Treated With Seroquel XR® (Quetiapine) and Other Atypical Antipsychotics.A 9-month, Observational, Multicentric Prospective Study.
Brief Title: Evaluating Subjective Well-being in Schizophrenic Patients Treated With quetiapineXR® and Other Atypical Antipsychotics
Acronym: Xperience
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Hans Eriksson, Medical Science Sr Director, AstraZeneca, Medical Science, Wilmington USA
Other Study IDs: NIS-NNL-SER-2008/1
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Last update posted 2010-10-27 (Estimated); Status verified 2010-10

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; remission; subjective well-being and effectiveness; Quality of Life
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
To evaluate the QOL (subjective effectiveness) in patients with schizophrenia, treated with atypical antipsychotics.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia
* Treatment with one atypical antipsychotic* (for a first/new episode or a switch of therapy) for at least 2 weeks and maximum 8 weeks prior to the first study visit.
* Patient takes an AAP according to local SPC and current medical practice
* The patient must be able to understand and comply with the study requirements as judged by the investigator, e.g. patient must be able to read and write

Exclusion Criteria:

* Treatment with an additional AAP or AP to the initial prescribed AAP within the 2-8 weeks before the patient is included in the study
* Since the use of clozapine is limited, due to, among other things, the risk for agranulocytosis, patients on treatment with this '2nd line'AAP are excluded.
* Previous enrolment or treatment in the present NIS
* Known allergy to the prescribed AAP or any of its substances

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with schizophrenia treated with atypical antipsychotics (AAPs) to stay in remission
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2008-04; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Subjective Wellbeing under Neuroleptics' SWN-K-score; Change from baseline of QoL assessed by the SWN-K after 9 months of treatment with atypical antipsychotics. | At baseline (Visit 1), and after ~3 months, ~6 months, ~9 months after V1, or at premature discontinuation

SECONDARY OUTCOMES:
Positive And Negative Syndrome Scale-PANSS-8score | At baseline (Visit 1), and after ~3 months, ~6 months, ~9 months after V1, or at premature discontinuation
Global Assessment of Functioning 'GAF' scale | At baseline (Visit 1), and after ~3 months, ~6 months, ~9 months after V1, or at premature discontinuation
Disease insight; G-12 item of PANSS | At baseline (Visit 1), and after ~3 months, ~6 months, ~9 months after V1, or at premature discontinuation

CONTACTS AND LOCATIONS:
Locations (37):
- Netherlands (37):
  - Research Site, Alphen
  - Research Site, Amersfoort
  - Research Site, Amstelveen
  - Research Site, Amsterdam
  - Research Site, Arnhem
  - Research Site, Bennebroek
  - Research Site, Boxmeer
  - Research Site, Breda
  - Research Site, Doetinchem
  - Research Site, Echt
  - Research Site, Enkhuizen
  - Research Site, Enschede
  - Research Site, Haarlem
  - Research Site, Halsteren
  - Research Site, Helmond
  - Research Site, Heythuysen
  - Research Site, Hoorn
  - Research Site, Kerkrade
  - Research Site, Kloetinge
  - Research Site, Leeuwarden
  - Research Site, Maastricht
  - Research Site, Nijmegen
  - Research Site, Oegstgeest
  - Research Site, Raalte
  - Research Site, Roermond
  - Research Site, Rotterdam
  - Research Site, Sluis
  - Research Site, Tiel
  - Research Site, Tilburg
  - Research Site, Utrecht
  - Research Site, Veenendaal
  - Research Site, Venray
  - Research Site, Vlaardingen
  - Research Site, Weert
  - Research Site, Zaandam
  - Research Site, Zoetermeer
  - Research Site, Zwolle